CLINICAL TRIAL: NCT03537560
Title: Detection of IDH2 Mutations and Monitoring Molecular Residual Disease in Patients With Acute Myeloid Leukemia
Brief Title: Detection of IDH2 Mutations and Monitoring Molecular Residual Disease in Patients With AML
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lee-Yung Shih, Professor, Chang Gung Memorial Hospital
Other Study IDs: 201700154B0
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Detection of IDH2 mutations in AML patients to define it incidence and correlation with clinical characteristics, relapse-free and overall survival.
2. Identify AML patients who are potential candidates for IDH2 inhibitor treatment.
3. Monitoring minimal residual disease (MRD) following therapy to evaluate its possible role in the strategy of MRD-directed therapy in the future in patients carrying IDH2 mutations at initial diagnosis.

DETAILED DESCRIPTION:
Isocitrate dehydrogenase 2 (IDH2) was found to be one of the recurrently mutated genes in acute myeloid leukemia, indicating its critical role in leukemogenesis. IDH2 mutations account for about 10%-20% of AML patients. IDH2 mutation is found to be associated with production of 2-HG, which interferes with histone methylation and DNA modification, results in partial block of myeloid cell differentiation. IDH inhibitors have shown in preclinical model to reverse differentiation blockage in tumor cells. The assessment of IDH2 inhibitors is ongoing with phase I/II clinical trials. The analysis of IDH2 mutation in AML patients will help to identify AML patients who might benefit from IDH inhibitor treatment.

Bone marrow samples from 300 adult patients (>20 years old) with newly diagnosed AML since 2014/1/1 and received standard chemotherapy in hospitals which has jointed Ministry of Health and Welfare AML program will be examined. The mononuclear cells are extracted from bone marrow samples at the initial diagnosis. The mutational analysis of exon 4 of IDH2 gene will be performed by PCR amplication followed by pyrosequencing to detect IDH2-R140 and R172 mutations and mutant levels. Follow-up samples of patients carrying IDH2 mutations at the time of achieving hematologic remission, subsequent samples during different time points including at least following two post-remission chemotherapy, at the end of therapy and every 3 months thereafter in the first year and then every 6 months up to 24 months, as well as at time of relapse, will be measured by LNA-quantitative real-time PCR with TaqMan probe assay to determine the changes of IDH2 mutant levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AML, age ≥ 20 years, and are willing to sign the informed consent

Exclusion Criteria:

* Not AML patients
* Patients diagnosed with AML but age < 20 years

Ages: 20 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with AML newly diagnosed and followed in Chang Gung Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Detection of IDH2 mutations | 1 month
  The mononuclear cells will be extracted from bone marrow samples at the initial diagnosis. The mutational analysis of exon 4 of IDH2 gene will be performed by PCR amplication followed by pyrosequencing to detect IDH2-R140 and R172 mutations and mutant levels.

SECONDARY OUTCOMES:
Follow-up detection of IDH2 mutations | 24 months
  Follow-up samples of patients carrying IDH2 mutations at the time of achieving hematologic remission, subsequent samples during different time points including at least following two post-remission chemotherapy, at the end of therapy and every 3 months thereafter in the first year and then every 6 months up to 24 months, as well as at time of relapse, will be measured by LNA-quantitative real-time PCR with TaqMan probe assay to determine the changes of IDH2 mutant levels.

CONTACTS AND LOCATIONS:
Overall Officials: Lee-Yung Shih, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital-Linkou, Taoyuan District, State, Taiwan